CLINICAL TRIAL: NCT02778789
Title: Non Randomized Parallel-group Clinical Study to Compare the Efficacy of Periarticular Bone Structure in Patients Treated With Either Tocilizumab or Tumor Necrosis Factor Blockers.
Brief Title: Comparing the Efficacy of Periarticular Bone Structure in Patients Treated With Either Tocilizumab or Tumor Necrosis Factor Blockers
Acronym: Re-Bone
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 1/4
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Adalimumab; Etanercept; golimumab; Certolizumab Pegol; Infliximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tocilizumab: Drug administration of Tocilizumab s.c. or i.v. depending on the preference of the patient and/or physician according to the label
  Interventions: Drug: Tocilizumab; Drug: TNF-alpha Inhibitor
- TNF-alpha Inhibitor: Drug administration s.c. or i.v. of the TNF-Alpha Inhibitor depending on the preference of the patient and/or physician according to the label
  Interventions: Drug: Tocilizumab; Drug: TNF-alpha Inhibitor

INTERVENTIONS:
Drug: Tocilizumab — Patients will be treated with either i.v. Tocilizumab every 4 weeks or s.c. Tocilizumab weekly according to the label
  Other Names: RoActemra
Drug: TNF-alpha Inhibitor — Patients will be treated with TNF-Inhibitors either i.v. or s.c. according to the label
  Other Names: Adalimumab, Etanercept, Golimumab, Certolizumab-Pegol, Infliximab

SUMMARY:
Comparing the structural effects of TNFi and tocilizumab on the periarticular bone by performing a comprehensive analysis of the periarticular bone changes in RA patients treated with either TNFi or tocilizumab in a longitudinal Setting, using high-resolution peripheral quantitative computed tomography (HR-pQCT), a very sensitive method for visualizing and quantifying bone microstructure in RA patients. Quantitatively assessing the changes of erosions volume, osteophytes size and the area of cortical fenestration in a group of TNFi-treated and a group of tocilizumab- treated RA patients.

DETAILED DESCRIPTION:
Inhibition of tumor necrosis factor alpha (TNF-α) and of interleukin- 6 receptor (IL-6R) emerged as highly effective cytokine blocking strategies in the treatment of rheumatoid arthritis (RA) in the last years. Both, inhibition of TNF-α (TNFi) and of the interleukin-6 receptor by tocilizumab ameliorate the signs and symptoms, reverse the elevated acute phase response and inhibit the progression of bone erosion in RA patients (1). Despite striking similarities with respect to their efficacy and safety in the treatment of RA, TNFi and tocilizumab are two entirely distinct approaches for targeting chronic inflammatory diseases in humans. This concept is highlighted by the differential response to TNFi and tocilizumab in other chronic inflammatory diseases such as psoriasis, psoriatic arthritis and spondyloarthritis, with clinical efficacy of the former but not the latter treatment modality (2). On the other hand, tocilizumab has a direct effect on the acute phase response and iron metabolism, which is not found with TNFi. Therefore, subtle differences may exist between TNFi and tocilizumab, which are relevant for the long-term treatment of RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Females and males with RA erosions in the wrist and/or MCP joints
* Must be aged ≥ 18 years at time of consent
* Stable treatment with conventional DMARDs of at least 3 months

Exclusion Criteria:

* Patients exposed to abatacept or rituximab in the last 12 months
* Patients receiving glucocorticoids over 5 mg prednisolone per day
* Patients who are younger than 18 years
* Pregnant or lactating females
* Patients having received an HR-pQCT examination during the last 6 months before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (ages over 18 years) with the diagnosis of RA will be screened for the presence of erosions by Routine procedure with HR-pQCT. In case of a positive scan showing the presence of erosion in the wrist or the MCP Joints and after the decision of the treatment (if either Tocilizumab or TNF-Inhibitor), patients will be enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09-30 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change in erosion volume in the HR-pQCT | 12 months

SECONDARY OUTCOMES:
Change in the Disease activity score 28 (DAS28) | 12months
Change in the Clinical Disease Activity Index (CDAI) | 12 months
Changes in the Simple Disease Activity Index (SDAI) | 12 months
Change in the Health Assessment Questionnaire (HAQ) | 12 months
Number of patients in Remission (DAS28 < 2.6) | 12 months
Number of patients in Low Disease Activity (DAS28 ≥ 2.6 und ≤ 3.2) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schett, Prof. Dr. univ., Principal Investigator — University of Erlangen-Nuremberg, Medical Department 3
Locations (1):
- University Erlangen-Nuremberg, Medical Department 3, Rheumatology & Immunology, Erlangen, Germany